CLINICAL TRIAL: NCT07341022
Title: HEMATOPOIETIC STEM CELL MOBILIZATION USING HIGH-DOSE PLERIXAFOR IN PATIENTS WITH SICKLE CELL DISEASE: A CONTROLLED PHASE I/II TRIAL.
Brief Title: STEM CELL MOBILIZATION WITH HIGH-DOSE PLERIXAFOR IN PATIENTS WITH SICKLE CELL DISEASE
Acronym: MobiSCD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MobiSCD Study
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; plerixafor; stem cell mobilization
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A: high-dose plerixafor (Experimental): 480 mcg/kg plerixafor
  Interventions: Drug: Plerixafor Dose Escalation

INTERVENTIONS:
Drug: Plerixafor Dose Escalation — Plerixafor will be administered as a single dose of 480 mcg/kg.

SUMMARY:
The objective of this study is to demonstrate whether high-dose plerixafor can effectively mobilize hematopoietic stem cells in patients with sickle cell disease. It will also learn about the safety of this drug in higher doses in these patients. The main questions it aims to answer are:

Does high-dose plerixafor mobilize enough hematopoietic stem cells? What medical problems do participants have when taking high-dose plerixafor?

Participants will:

Undergo transfusion Take high-dose plerixafor Be submitted to stem cell collection by apheresis Visit the clinic 10 days after the procedure Be contacted by the research team 30 days after the procedure.

DETAILED DESCRIPTION:
Sickle cell disease (SCD), the most common monogenic disorder in the world, is currently considered a global public health problem, which underscores the need to develop curative therapies for this condition. Gene therapy has been emerging as a safe and effective curative therapeutic strategy, with the advantage of using autologous hematopoietic progenitor cells (HPCs) that are collected from the patient, edited in the laboratory, and reinfused-a process known as ex vivo gene therapy. However, mobilizing and collecting HPCs in this population is challenging, both due to disease-related factors such as bone marrow inflammation, necrosis, and ineffective erythropoiesis, and because the quantity of HPCs required for gene therapy protocols is very high. Since the use of granulocyte colony-stimulating factor (G-CSF) is contraindicated in SCD, the CXCR4 inhibitor plerixafor has been validated in this population as a safe drug, although with variable effectiveness. In healthy volunteers, plerixafor has been tested at twice the usual dose, with a significant increase in mobilization efficacy. However, in the context of sickle cell disease, and even in other diseases, this approach has never been tested. Additionally, although plerixafor is already approved for commercial use for other conditions in Brazil, it has never been tested in patients with SCD in our country, whose genetic background is more ethnically admixed compared to populations in high-income countries. This project aims to assess the efficacy and safety of plerixafor in a population of Brazilian patients with SCD. To do so, 12 patients will be enrolled using an adaptive design model that will include 3 patients at a time. The primary endpoint will be the proportion of patients who achieve a CD34+ cell count after HPC collection > 5×10⁶/kg of body weight following a single dose of plerixafor at 480 mcg/kg. Secondary endpoints will evaluate safety, efficacy, preservation of cell potency, and a preliminary cost-effectiveness analysis. This study not only introduces an unprecedented approach but also validates findings from other studies in a genetically diverse population. Moreover, it brings to Brazil the expertise necessary for HPC mobilization in SCD, an essential step for the success of future clinical gene therapy protocols to be implemented based on ongoing preclinical studies in the country, with potential for incorporation into the Brazilian Unified Health System (SUS).

ELIGIBILITY:
Inclusion Criteria:

Patients with sickle cell disease 18 to 25 years old At least one allogeneic HSCT indication followin the Brazilian Bone Marrow Transplant Society (SIMÕES et al., [s.d.]) ECOG/ Karnofsky/Lansky scores > 80 Hemoglobin > 7 g/dL, WBC counts > 3000/mm3, neutrophil counts > 1500/mm3, platelet counts > 150000/mm3 No evidence of severe hepatic disfunction, defined as aspartate aminotransferase and alanine aminotransferase < 5 times ULN or bilirubin < 2,5 times ULN No evidence of renal disfunction, defined as creatinine <1,5 mg/dL ou GFR> 60 mL/min LVEF > 40% and no signals of pulmonary hypertension Negative serologies for HIV, HBV, HCV, syphilis, Chagas disease or HTLV Being able to undergo partial exchange transfusion to lower HbS <30% within one week before CD34+ mobilization and collection No pregnancy or breastfeeding; acceptance to use two contraceptive methods during the study.

Exclusion Criteria:

Emergency room admission or hospitalization in the past 14 days prior to first dose of study drug Major surgery in the past 30 days prior to first dose of study drug Active and painful splenomegaly or splenomegaly (size greater than upper limit of normal on examination).

Participant who, by medical history, requires rare donor registry RBC units for transfusion, or is unable to receive routine transfusion. Eligible study participants must have undergone prior work-up for the presence of red cell alloantibodies and confirmation of available compatible blood product support Known allergy to or contraindication for motixafortide administration, or medications routinely administered during apheresis Participant who has had a prior autologous or allogeneic transplantation, inclusive of gene therapy Active viral, bacterial, fungal, or parasitic infection. History of cancer, excluding squamous carcinoma of the skin and cervical carcinoma in situ.

Participant who has received experimental therapy within 4 weeks prior to providing informed consent Poorly controlled diabetes mellitus, as assessed by the Investigator Concomitant treatment with alternative investigational agent unable to be held for 30 days Unwillingness to use a highly effective method of contraception for 1 month after motixafortide Pregnancy Inability or unwillingness of research participant or legal guardian/ representative to give written informed consent.

Inability or unwillingness of research participant to hold hydroxyurea for 30 days prior to first dose of study drug

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
CD34⁺ cell count | 0 days
  Proportion of patients who achieve a CD34⁺ cell count > 5 × 10⁶/kg body weight after HSC collection using plerixafor at a dose of 480 µg/kg

IPD SHARING:
Plan to Share IPD: No